CLINICAL TRIAL: NCT00386529
Title: A Multi-center, Double-Blind Randomized, Cross-over, Active-control, Comparative Clinical Study to Evaluate the Administration Time-dependent Antihypertensive Effects of Low Dose Aspirin in Well-Controlled Hypertensive Patients (Phase IV)
Brief Title: Administration Time-dependent Antihypertensive Effects of Low Dose Aspirin in Well-controlled Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Kyungpook National University Hospital (Other); The Catholic University of Korea (Other); Cheil General Hospital and Women's Healthcare Center (Other); Inje University (Other); Keimyung University (Other); Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Yeungnam University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AST-HT-01
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Well-controlled Hypertension
Keywords: low dose aspirin; Hypertension; administration time dependent effect
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aspirin enteric coated pellests 100mg

SUMMARY:
The purpose of this study is to evaluate the influence of aspirin on blood pressure in well-controlled hypertensive patients who receive low dose aspirin at different times of the day

DETAILED DESCRIPTION:
Recent studies showed that low dose aspirin exerts a significant administration time-dependent effect on blood pressure in previously untreated hypertensive patients. However, this effect has not been confirmed in patients taking low-dose aspirin in combination with antihypertensive medications. A multi-center, double-blind randomized, cross-over, active-control, comparative clinical study will be conducted to evaluate the influence of aspirin on blood pressure in well-controlled hypertensive patients who receive low dose aspirin at different times of the day.

Approximately 192 patients will be enrolled over 4 months in 8 centers nationwide.

After placebo run-in period, all subjects will be randomized into one of the following 3 groups.

Group I & II will take low dose aspirin for treatment period (for first and second 12 weeks)on awakening or before bed time. Group III will take placebo for treatment period.

After first 12 weeks' treatment period, the subjects will be informed whether she/he belongs to Group III. This will be done without breaking the double blinding in the other 2 groups.

The primary objective will be the evaluation of the influence of aspirin on blood pressure in well-controlled hypertensive patients who receive low dose aspirin at different times of the day.

The secondary objectives will be 1) comparison of the administration time-dependent effects of low dose aspirin on blood pressure between dipper and non-dipper patients and 2) the evaluation of the effects of low dose aspirin in Korean hypertensive patients.

A sub-study will be conducted in 3 centers to evaluate the effect of aspirin on endothelial function in patients with well-controlled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age : 30 - 70 (inclusive)
* Essential hypertension without complication
* Well-controlled blood pressure over 3 months with same antihypertensive medication without changes in dose and frequency
* Averages of two consecutive sitting diastolic and systolic blood pressures are <90 mmHg and <140 mmHg, respectively at screening and visit 1
* Differences in sitting diastolic and systolic blood pressures between screening and visit 1 are 10 mmHg and 20 mmHg, respectively.
* Willing and able to give informed consent

Exclusion Criteria:

* patients with sitting diastolic blood pressure < 70 mmHg
* patients with secondary or malignant hypertension
* patients with complication or high risk of complication
* proven coronary artery or peripheral vascular diseases
* Framingham CHD Risk Score (10 years) 20
* Fasting blood glucose 110 mg/dl
* Hyperlipidemia under treatment or treatment required
* patients with myocardial infarction or severe cerebrovascular disorder in last 6 months
* patients with chronic renal insufficiency
* patients with unstable angina
* patients with severe left ventricular abnormalities or valvular defect
* patients with bradycardia(pulse rate < 50 times/min) or chronic tachycardia (pulse rate 100 times/min), second degree AV-block
* SGOT, SGPT> 2.5 times upper limit range or serum creatinine > 1.5 times upper limit range
* patients with unresolved malignant tumor or systemic infection
* lactating or pregnant females or females of childbearing potential who do not undergo hysterectomy or are not willing to use "effective" method of contraception.
* known hypersensitivities to the investigational drug
* patients judged to have alcohol or other drug abuse by the investigator
* patients who takes contraindicated drug at study entry (visit 1) or needs to contraindicated drug throughout the study period(if judged by the investigator not to influence on the study due to the temporal administration etc.)
* patients judged to be inappropriate for this study be the investigator
* patients with gastrointestinal troubles to NSAIDs

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2006-09; Primary Completion 2007-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
the changes in diastolic blood pressure

SECONDARY OUTCOMES:
the changes in systolic blood pressure
the trend in home blood pressure for medication
the comparison of the changes in systolic and diastolic pressure in dipper and non-dipper patients

CONTACTS AND LOCATIONS:
Overall Officials: Shung Chull Chae, Professor, Study Chair — Kyungpook National University Hospital; Dong Ju Choi, Professor, Principal Investigator — Seoul National University Bundang Hospital; Dong Su Kim, Professor, Principal Investigator — Inje University; Jeong Bae Park, Professor, Principal Investigator — Cheil General Hospital and Women's Healthcare Center; Nam Sik Chung, Professor, Principal Investigator — Severance Hospital; Sang Hong Baek, Professor, Principal Investigator — The Catholic University of Korea; Chang Wook Nam, Professor, Principal Investigator — Keimyung University Dongsan Medical Center; Young Jo Kim, Professor, Principal Investigator — Yeungnam University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

REFERENCES:
- [Result] Avanzini F, Palumbo G, Alli C, Roncaglioni MC, Ronchi E, Cristofari M, Capra A, Rossi S, Nosotti L, Costantini C, Pietrofeso R. Effects of low-dose aspirin on clinic and ambulatory blood pressure in treated hypertensive patients. Collaborative Group of the Primary Prevention Project (PPP)--Hypertension study. Am J Hypertens. 2000 Jun;13(6 Pt 1):611-6. doi: 10.1016/s0895-7061(00)00231-4. PMID 10912743
- [Result] Magen E, Viskoper JR, Mishal J, Priluk R, London D, Yosefy C. Effects of low-dose aspirin on blood pressure and endothelial function of treated hypertensive hypercholesterolaemic subjects. J Hum Hypertens. 2005 Sep;19(9):667-73. doi: 10.1038/sj.jhh.1001910. PMID 16034448
- [Result] Hermida RC, Fernandez JR, Ayala DE, Mojon A, Iglesias M. Influence of aspirin usage on blood pressure: dose and administration-time dependencies. Chronobiol Int. 1997 Nov;14(6):619-37. doi: 10.3109/07420529709001452. PMID 9360028
- [Result] Hermida RC, Ayala DE, Iglesias M. Administration time-dependent influence of aspirin on blood pressure in pregnant women. Hypertension. 2003 Mar;41(3 Pt 2):651-6. doi: 10.1161/01.HYP.0000047876.63997.EE. Epub 2002 Dec 9. PMID 12623974
- [Result] Hypertension 2005;46[part2]:1060-1068